CLINICAL TRIAL: NCT06815549
Title: An Open Clinical Trial of the Safety and Efficacy of the Drug Fluorothiazinone, 300 Mg Tablets (Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation) with the Participation of Adult Patients with Chronic Bacterial Cystitis"
Brief Title: An Open Clinical Trial of the Safety and Efficacy of the Drug Fluorothiazinone, 300 Mg Tablets with the Participation of Adult Patients with Chronic Bacterial Cystitis"
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-FT-2024
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: P. Aeruginosa; Baumannii; Klebsiella Pneumonia; E.coli Infections; Enterococcus Faecalis Infection; Chronic Bacterial Cystitis
MeSH Terms: interventions — Tablets; Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: Fluorothiazinone, tablets 300 mg (Experimental): Treatment arm patients will receive Fluorothiazinone, tablets 300 mg at a dose 1200 mg/day (2 tablets twice a day) for 14 days.
  Interventions: Drug: Fluorothiazinone, tablets 300 mg
- Comparator: Nitrofurantoin (Active Comparator): Comparison arm patients will receive Nitrofurantoin in accordance with the instructions for medical use.
  Interventions: Drug: Nitrofurantoin 100 MG

INTERVENTIONS:
Drug: Fluorothiazinone, tablets 300 mg — patients will receive Fluorothiazinone, tablets 300 mg at a dose 1200 mg/day (2 tablets twice a day) for 14 days
  Arms: Drug: Fluorothiazinone, tablets 300 mg
Drug: Nitrofurantoin 100 MG — Comparison arm patients will receive Nitrofurantoin in accordance with the instructions for medical use.
  Arms: Comparator: Nitrofurantoin

SUMMARY:
This study is designed to evaluate the safety, clinical efficacy and antibacterial activity of the drug Fluorothiazinone, 300 mg tablets, (Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation) in the mode of antibacterial monotherapy with the participation of adult patients with chronic bacterial cystitis.

The main objectives of this study are:

1. To evaluate the safety of the use of the drug Fluorothiazinone according to the indicators

   1. adverse events/reactions;
   2. serious adverse events/reactions;
   3. deviations from clinical and laboratory parameters.
2. To evaluate the therapy effectiveness:

   1. clinical cure - complete resolution or improvement of the signs and symptoms of chronic cystitis that were present at baseline and the absence of new symptoms requiring antimicrobial therapy on days 7, 14 and 28 after the start of therapy;
   2. the timing of the disappearance of symptoms according to the patient's subjective feelings;
   3. microbiological response when comparing pre-treatment and post-treatment cultures;
   4. changes on VAS (visual analogue scale) for pain intensity determination;
   5. changes on PUF (Pelvic pain and urgency/frequency patient symptom scale) for assessing symptoms by patients;
   6. changes on ACSS (acute cystitis symptom scale);
   7. development of relapses within 90 days after the start of therapy.
3. To collect clinical isolates of pathogens for molecular genetic analysis. The identification of DNA and the determination of the bacterial genotype will allow us to assess the microbiological outcomes such as relapse or reinfection.
4. To determine the sensitivity of the obtained isolates to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written consent to participate in the study in accordance with the current legislation.
2. The ability to understand the requirements for the study participants, the willingness to follow the procedures according to the Study Protocol.
3. Female Patients, at least 18 years old.
4. Ambulatory treatment, absence of indications for emergency hospitalization during the period of inclusion in the study for the infection under study.
5. Bacterial cystitis, a history of chronic recurrent bladder infection.
6. The presence of symptoms characteristic of exacerbation of chronic cystitis: pain syndrome (pain in the lower abdomen, when urinating), dysuric symptoms (frequent urination, pain or burning when urinating, imperative urge to urinate, feeling of incomplete emptying of the bladder). 6 points or higher when assessing the characteristic symptoms on the ACSS scale.
7. Consent of patients with preserved reproductive potential to use effective methods of contraception using one of the following methods: abstinence, intrauterine device, oral/ injectable contraceptive, subcutaneous implant or double barrier method (condom with local contraceptive) for the period of participation in the study.
8. Negative pregnancy test result before randomization for female patients with preserved reproductive potential.

Exclusion Criteria:

1. Inability to read in Russian; inability or unwillingness to understand the essence of the research. Any other conditions that limit the validity of obtaining informed consent or may affect the volunteer's ability to participate in the study.
2. Participation in any other study in the last 90 days;
3. Presence of an infection of another organ other than a bladder infection, such as endocarditis, osteomyelitis, abscess, meningitis, pneumonia, etc.
4. Symptoms requiring hospitalization (macrohematuria, concomitant diseases that complicate the course of the disease).
5. Cystocele of 3-4 degrees.
6. Treatment with Nitrofurantoin for 30 days before randomization.
7. Mental illness (registered by a psychiatrist according to medical records).
8. Treatment with hormonal drugs (with the exception of hormonal contraceptives, hormone replacement therapy, topical medications) for the last 10 days.
9. Autoimmune diseases or systemic connective tissue diseases in the anamnesis, requiring the appointment of immunosuppressive therapy.
10. Recipients of solid organs or tissues (bone marrow or peripheral blood stem cells).
11. Taking immunosuppressive drugs and/or immunomodulators for 6 months prior to the start of the study.
12. The presence of congenital or acquired immunodeficiency (AIDS, etc. according to medical history).
13. History of malignant neoplasms, with the exception of basal cell or squamous cell epithelial carcinomas of the skin, which were removed without signs of metastasis more than 3 years ago.
14. Blood donation (450 ml or more of blood or plasma) less than 2 months before the start of the study.
15. Planned hospitalization and / or surgical intervention during the period of participation in the study, as well as 4 weeks before the expected date of drug administration.
16. The presence of a concomitant disease that may affect the evaluation of the results of the study or which, in the opinion of the investigator, will not allow the patient to participate in the study or may affect the conduct of the study and / or its results (including the assessment of safety parameters), any conditions that, in the opinion of the medical investigator, may be a contraindication to participating in the study.
17. Pregnancy or breast-feeding.
18. Taking any long-acting systemic antibiotic (i.e., with a frequency of administration no more than once a day) for less than 12 hours before randomization.
19. The need at the time of randomization for additional systemic antimicrobial therapy (including antibacterial, antifungal therapy) other than treatment with the investigational drug, with the exception of a single oral administration of any antifungal drug for the treatment of vaginal candidiasis.
20. Lactose intolerance, lactase deficiency or glucose-galactose malabsorption, allergy to the components of the studied drug / reference drug in the anamnesis.
21. Contraindications to the use of Nitrofurantoin (severe renal excretory function disorders, renal insufficiency, oliguria, glucose-6-phosphate dehydrogenase deficiency, hypersensitivity to Nitrofurantoin, stage II-III heart failure, liver cirrhosis, chronic hepatitis, acute porphyria).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs | Within 90 days after administration of the drug.
  Occurrence of adverse events/reactions.
SAEs | Within 90 days after administration of the drug.
  Occurrence of serious adverse events/reactions.
Complete resolution or improvement of the signs and symptoms of chronic cystitis | 7th, 14th and 28th days after the start of therapy.
  Complete resolution or improvement of the signs and symptoms of chronic cystitis that were present at baseline, and the absence of new symptoms, that require further antimicrobial therapy.
Relapse | Within 90 days from the start of therapy.
  Relapse of chronical bacterial cystitis monitoring.

IPD SHARING:
Plan to Share IPD: No